CLINICAL TRIAL: NCT06710431
Title: A Double-blind, Placebo-controlled, Phase IIA Human Laboratory Study of the Safety and Exploratory Efficacy of Oral AFA-281 in Patients with Alcohol Use Disorder
Brief Title: A Study of the Safety and Exploratory Efficacy of Oral AFA-281 in Patients with Alcohol Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Afasci Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AFA-281-304
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Alcohol Abuse; Alcohol Abuse/addiction; Anxiety; Pain Threshold; Depression Disorders; Sleep Disorder
Keywords: AFA-281; alcohol abuse; alcohol; depression; pain threshold; sleep disorder; anxiety
MeSH Terms: conditions — Alcoholism; Behavior, Addictive; Anxiety Disorders; Sleep Wake Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- AFA-281 placebo control (Placebo Comparator): AFA-281 placebo control group
  Interventions: Drug: AFA-281
- Low dose of AFA-281 (Active Comparator): AFA-281 at 60 mg per day
  Interventions: Drug: AFA-281
- High dose AFA-281 (Active Comparator): AFA-281 at 120 mg per day
  Interventions: Drug: AFA-281

INTERVENTIONS:
Drug: AFA-281 — AFA-281

SUMMARY:
This study will evaluate the safety and exploratory efficacy of AFA-281 in patients with Alcohol use disorder on cravings, subjective response to alcohol, pain thresholds, anxiety, depression, and sleep.

DETAILED DESCRIPTION:
This study will determine the safety, tolerability, and exploratory efficacy of AFA-281. This study is a randomized, double-blind, placebo-controlled, human laboratory study of 36 community-based, non-treatment-seeking male and female individuals with current (i.e., past month) moderate-to-severe AUD (DSM-5). This study will be conducted by Dr. Lara Ray at UCLA. The total study duration is approximately 42 days including a 2-week screening period. Eligible participants will be randomized into one of three cohorts: 60 mg AFA-281, 120 mg AFA-281, or Placebo. Participants will start at a lower dose and increase the dose over 2 weeks then continue to maintain the dose for an additional 2 weeks. In week 4, participants will complete 7 daily visits to complete assessments and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 21 and 65
2. Must voluntarily sign and date each informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures.
3. Meet current (i.e., past 12 months) DSM-5 diagnostic criteria for moderate or severe AUD
4. Report drinking at least 28 drinks per week if male, 21 drinks per week if female, in the 28 days prior to consent.
5. Must be surgically sterile (vasectomy, tubal ligation, or hysterectomy) or agree to be sexually inactive or agree to use a barrier method of birth control (i.e., condom) from the start of screening until study completion, and agree to refrain from donating sperm for 90 days after study drug administration.

Exclusion Criteria:

1. Current treatment for alcohol use or a history of treatment in the 30 days before enrollment or treatment seeking
2. Current (last 12 months) DSM-5 diagnosis of dependence on any psychoactive substances other than nicotine
3. Current DSM-5 diagnosis of substance use disorder for any substance other than alcohol and nicotine
4. Lifetime DSM-5 diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder
5. Current DSM-5 major depressive disorder with suicidal ideation
6. Positive urine screen for narcotics, amphetamines, or sedative hypnotics
7. Clinically significant alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised
8. Pregnancy, nursing, or refusal to use reliable method of birth control if female
9. History of significant sensitivity to any drug.
10. Has a clinically significant abnormal ECG or an ECG with a QTc interval corrected for heart rate using the Fridericia formula (QTcF) > 430 ms.
11. History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, endocrine, dermatological, metabolic or psychiatric disease or disorder, or any uncontrolled medical illness.
12. Has an estimated creatinine clearance (CrCl) outside of normal range.
13. History of head trauma with loss of consciousness, seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
14. History of gastric surgery, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH, or absorption.
15. Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or HIV antibodies (HIV Ab). Negative HIV status will be confirmed at Screening and the results will be maintained confidentially by the study site.
16. Liver enzymes AST, ALT, or GGT ≥ 3 times upper normal limit.
17. Positive urine drug screen for drugs of abuse at Screening or Day -1.
18. Receipt of any drug by injection within 30 days prior to study drug administration.
19. A clinically notable vital sign abnormality including a history of syncopal or near syncopal events following abrupt change in posture.
20. Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration.
21. Pregnant or nursing women.
22. Receipt of any investigational products within 6 weeks prior to study drug administration.
23. Current enrollment in another clinical study.
24. Previous enrollment in this study.
25. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to participate in the AFA-281 Phase I1a Study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Cue-induced alcohol craving | predose and weekly through Week 4
  Questionnaire measures the level of alcohol craving
Stress-induced alcohol craving | predose and weekly through Week 4
  Alcohol urge questionnaire after stressful stimuli
Subjective response to alcohol | predose and weekly through Week 4
  Biphasic alcohol effects scale and profile of negative mood states
Pain assessments | predose and weekly through Week 4
  Latency to first feel pain and pain intensity scoring using the McGill Pain Questionnaire
Safety and tolerability assessment | Predose and Daily
  Daily questions via CAROMA system

SECONDARY OUTCOMES:
Daily diary report | predose and weekly through Week 4
  Examination of clinically relevant phenotypes by daily diary reports of alcohol use, alcohol craving, anxiety, depression, subjective pain and sleep

CONTACTS AND LOCATIONS:
Overall Officials: Lara Ray, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided